CLINICAL TRIAL: NCT01306682
Title: Trivalent Influenza Vaccine in HIV-infected Pregnant Women and Kinetics of Transplacental Anti-influenza Antibody Transfer and Persistence in Young Infants: A Randomized Controlled Phase II Trial Evaluating Safety and Immunogenicity
Brief Title: Influenza Vaccination of HIV Infected Pregnant Women: Safety and Immunogenicity
Acronym: MatfluHIVpos
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Emory University (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Michelle Groome, Medical officer, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Maternal_flu_HIVpos_101107
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; vaxigrip; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent Influenza vaccine (Active Comparator): 0.5ml of TIV will be administered into deltoid muscle of non dominant arm
  Interventions: Biological: Trivalent influenza vaccine
- Normal saline (Placebo Comparator): 0.5ml of normal saline administered into deltoid muscle of non dominant arm
  Interventions: Biological: Normal saline

INTERVENTIONS:
Biological: Trivalent influenza vaccine — 0.5 ml of trivalent influenza vaccine administered into deltoid muscle of non dominant arm
  Other Names: Vaxigrip
  Arms: Trivalent Influenza vaccine
Biological: Normal saline — 0.5ml normal saline administered into deltoid muscle of non dominant arm
  Other Names: NaCl
  Arms: Normal saline

SUMMARY:
This randomized, placebo controlled trial will evaluate the safety and immunogenicity of Trivalent Influenza Vaccine (TIV) in HIV-infected pregnant women, dynamics of transplacental anti-influenza antibody transfer to their newborns and kinetics thereof during early infancy.

DETAILED DESCRIPTION:
Determining the contribution of influenza to early childhood morbidity and mortality in sub-Saharan Africa and the potential to prevent influenza disease through vaccination may contribute to reducing childhood deaths; since influenza illness is a vaccine preventable disease for which vaccines are developed, licensed and available at reasonable cost. Unfortunately, infants at highest risk for serious disease are those under 6 months of age, for whom trivalent inactivated influenza vaccine (TIV) is poorly immunogenic and not licensed. As pregnant women also have an increased risk of serious illness (3.3-5.5 fold for hospitalization for influenza-associated acute cardio-respiratory illness) from influenza infection, one strategy to prevent the complications of influenza in pregnant women and young infants is through maternal TIV immunization, which is recommended by the WHO. This could result in direct protection of the women and protection of the young infant consequent to transplacental transfer of TIV induced antibody.

Barriers to administration of vaccines during pregnancy including lack of information on effectiveness and concerns about safety probably explain the virtual non-existent use of TIV in pregnant women from low-middle income countries, including South Africa.

The immunogenicity and efficacy of TIV in HIV-infected adults was only recently documented in an African setting. A placebo-controlled, community-based randomized, placebo controlled trial, conducted in South Africa reported that TIV was associated with a 75% reduction in influenza-confirmed illness. The results of the study also confirmed the safety of TIV among African HIV-infected adults. The study, however, only included 7 women who were pregnant. In addition to no differences in solicited adverse event rates, there was also no difference in either CD4+ cell count changes or HIV viral control in those on antiretroviral treatment between TIV vaccinees compared to placebo recipients. This allayed previous concerns regarding the potential negative effect of TIV which centered around the observed transient increase in HIV-1 viral load, even in HIV infected individuals on ART and who were virologically suppressed (viral load <400 copies/ml). Decreases in CD4+ lymphocyte counts have also been observed in HIV-infected individuals post TIV vaccination. These changes, however, even in past studies were infrequent (4-18%) and resolved at later time-points and were considered to be clinically non-significant.

Only recently has data become available from Bangladesh in which the benefit of maternal TIV vaccination was demonstrated by a 63% (95%CI 5 to 85) reduction in laboratory-confirmed influenza illness in infants under 24 weeks of age in children born to mothers vaccinated with TIV and a 36% reduction in clinical illness in vaccinated mothers. There has, however, not been any study on the effectiveness of maternal immunization with TIV on influenza- associated morbidity and mortality either in the mothers or infants in African settings.

Despite the encouraging results on maternal immunization from Bangladesh, and the preliminary data supporting that TIV is efficacious mainly in HIV-infected non-pregnant adults, further data are needed to advocate for routine use of TIV during pregnancy in settings with a high prevalence of HIV. Reasons for this include that the impact of maternal HIV on the kinetics of TIV induced transplacental antibody transfer cannot be derived from available data. This is important as the primary focus of this proposal, and major potential public health benefit of maternal TIV vaccination, is targeted at protection of young infants. HIV infection is known to decrease placental integrity and lower antibody levels in the fetus and newborn. Furthermore, maternal hypergamma-globulinemia that is characteristic of HIV-infection may be associated with decreased neonatal antibody levels. This paradox is explained by the limited number of placental antibody receptors, resulting in IgG antibodies competing for available receptors and thereby decreasing vaccine-specific antibody transport. Preterm birth increases with HIV, chronic maternal disease or malnutrition. Transfer of maternal antibody which is gestational age dependant, may be more affected by maternal immunization in sub-Saharan Africa where these conditions are common.

The overall aim of this project is to evaluate the safety and immunogenicity of TIV vaccination of HIV-infected pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age > 18 years to < 39 years.
* Gestational age ≥ 20 weeks to < 34 weeks documented by the approximate date of the last menstrual period and corroborated by physical exam.
* Documented to be HIV-infected on two assays prior to study-enrollment.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of study.

Exclusion Criteria

* In HIV-infected women features of WHO clinical category 3 or 4 of AIDS at the time of enrollment.
* Receipt of TIV, other than through the study, during the current influenza season documented by medical history or record.
* Receipt of any live licensed vaccine ≤ 28 days or inactivated licensed vaccine ≤ 14 days prior to study-vaccine.
* Receipt of a non-licensed agent (vaccine, drug, biologic, device, blood product, or medication) ≤ 28 days prior to vaccination in this study, or expects to receive another non-licensed agent before delivery unless study approval is obtained.
* Any significant (in the opinion of the site investigator) acute illness and/or oral temperature greater than or equal to 38 degrees C ≤ 24 hours prior to study entry.
* Use of anti-cancer systemic chemotherapy or radiation therapy ≤ 48 weeks of study enrollment, or has immunosuppression as a result of an underlying illness or treatment.
* Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) ≤ 12 weeks of study entry, or high-dose inhaled steroids (> 800 mcg/day of beclomethasone dipropionate or equivalent) ≤ 12 weeks before study entry (nasal and topical steroids are allowed).
* Receipt of corticosteroids for preterm labor ≤ 14 days before study entry.(ix) Receipt of immunoglobulin or other blood products (with exception of Rho D immune globulin) ≤ 12 weeks prior to enrollment in this study or is scheduled to receive immunoglobulin or other blood products (with the exception of Rho D immune globulin) during pregnancy or for the first 24 weeks after delivery.
* Receipt of IL2, IFN, GMCSF or other immune mediators ≤ 12 weeks before enrollment.
* Uncontrolled major psychiatric disorder.
* History of a severe adverse reaction to previous TIV.
* Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Pregnancy complications (in the current pregnancy) such as pre-term labor, hypertension (systolic blood pressure ≥ 140 and/or diastolic blood pressure ≥ 90 mm Hg) or pre-eclampsia

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Humoral immune responses to influenza strains in the vaccine will be measured to assess the immunogenicity of TIV in HIV-infected pregnant women vaccinated between 20-34 weeks of gestational age | 1 month post vaccination, delivery (+7 days), 24 weeks post delivery
  Humoral immunity will be measured by hemagglutination inhibition (HAI) assay. Blood will be collected at enrolment (pre-vaccination), one month post vaccination, delivery (+7 days) and 24 weeks post delivery. Humoral immune response definitions: HAI titers < 1:10 = seronegative; ≥ 1:10 = seropositive; > 1:40 = protected against influenza; Response to TIV = serconversion (from <1:10 to ≥1:10) and/or 4-fold increase of HAI titers.
The proportion of newborns born to HIV-infected mothers with hemagglutination inhibition (HAI) antibody titers of ≥1:40 to TIV strain will be determined and compared to newborns born to TIV-vaccinated HIV-uninfected women (parallel trial) | Delivery (+7 days)
  Determine the proportion of newborns with hemagglutination inhibition (HAI) antibody titers of ≥1:40 to each of the three TIV strains born to HIV-infected mothers and compared to newborns born to TIV-vaccinated HIV-uninfected women

SECONDARY OUTCOMES:
Hemagglutinin (HA) antibody measurements in blood taken from mother and infants up to 24 weeks post delivery will be used to assess dynamics and kinetics of transplacentally acquired antibodies | 24 weeks post partum
  Hemagglutinin (HA) antibody measurements in blood taken from mother at birth and infants at birth, 8,16 and 24 weeks post delivery will be used to assess dynamics and kinetics of transplacentally acquired antibodies
The number of laboratory-confirmed or clinical influenza like illness cases in infants born to HIV infected mothers who received TIV or placebo will be used to determine efficacy of TIV vaccination of pregnant women against ILI in their infants | 24 weeks of age
  All infants (up to 24 weeks of age) born to women enrolled on trial will be assessed by study staff if they have any signs or symptoms (including fever, hospitalisation, apnea, cough, nasal catarrh/ congenstion, tachypnea) which could indicate influenza like illness. Nasopharyngeal aspirate samples collected at illness visits will be processed for viruses using real time reverse transcriptase-polymerase chain reaction (rRTPCR) assays.
The number of laboratory-confirmed influenza illnesses and clinical ILI cases in maternal participants during pregnancy and for 24 weeks post-partum will be used to assess efficacy of TIV against laboratory confirmed and clinical ILI | 24 weeks
  All maternal participants with signs and/ or symptoms of influenza like illness (ILI) will have nasopharyngeal and oropharyngeal swabs collected at illness visits and processed by rRTPCR assays. Participants from whom influenza virus is isolated at illness visits will be included in analysis to evaluate the efficacy of TIV against laboratory-confirmed influenza illness in mothers during pregnancy and until 24 weeks post-partum. Participants with no influenza isolated will be included in analysis of clinical ILI.
Cell-mediated immune (CMI) responses to influenza strains in the vaccine will be measured to define CMI responses to TIV in HIV infected pregnant women | 1 month post vaccination
  Cell mediated immunity will be measured by ELISPOT response to TIV. Blood will be collected at enrollment (pre-vaccination) and one month post vaccination
CD4+ and HIV-viral load will be measured at baseline and one-month post vaccination to evaluate effect of TIV. | 1 month post vaccination
  Evaluate the effect of TIV on CD4+ and HIV-viral load changes comparing baseline levels to one-month post vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Study Chair — University of Witwatersrand, South Africa; Keith P Klugman, MD, PhD, Study Director — Emory University; Adriana Weinberg, PhD, Study Director — University of Colorado, Denver
Locations (1):
- RMPRU, Chris Hani Baragwanath Hospital, Soweto, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Motsoeneng BM, Dhar N, Nunes MC, Krammer F, Madhi SA, Moore PL, Richardson SI. Hemagglutinin Stalk-Specific Fc-Mediated Functions Are Associated With Protection Against Influenza Illness After Seasonal Influenza Vaccination. J Infect Dis. 2024 Dec 16;230(6):1329-1336. doi: 10.1093/infdis/jiae241. PMID 38743692
- [Derived] Madhi SA, Cutland CL, Downs S, Jones S, van Niekerk N, Simoes EAF, Nunes MC. Burden of Respiratory Syncytial Virus Infection in South African Human Immunodeficiency Virus (HIV)-Infected and HIV-Uninfected Pregnant and Postpartum Women: A Longitudinal Cohort Study. Clin Infect Dis. 2018 May 17;66(11):1658-1665. doi: 10.1093/cid/cix1088. PMID 29253090
- [Derived] Madhi SA, Nunes MC, Weinberg A, Kuwanda L, Hugo A, Jones S, van Niekerk N, Ortiz JR, Neuzil KM, Klugman KP, Simoes EAF, Cutland CL; Maternal Flu Trial (Matflu) Team. Contribution of Serologic Assays in the Evaluation of Influenza Virus Infection Rates and Vaccine Efficacy in Pregnant Women: Report From Randomized Controlled Trials. Clin Infect Dis. 2017 Jun 15;64(12):1773-1779. doi: 10.1093/cid/cix241. PMID 28369198
- [Derived] Madhi SA, Cutland CL, Kuwanda L, Weinberg A, Hugo A, Jones S, Adrian PV, van Niekerk N, Treurnicht F, Ortiz JR, Venter M, Violari A, Neuzil KM, Simoes EA, Klugman KP, Nunes MC; Maternal Flu Trial (Matflu) Team. Influenza vaccination of pregnant women and protection of their infants. N Engl J Med. 2014 Sep 4;371(10):918-31. doi: 10.1056/NEJMoa1401480. PMID 25184864